CLINICAL TRIAL: NCT03285737
Title: Whey Protein Intake in the Amelioration of Skeletal Muscle Quantity and Function During Inactivity in Older Adults
Brief Title: Protein Intake and Step Reduction in Older Adults
Acronym: DRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: National Dairy Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HIREB 0574
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2017-09

CONDITIONS: Aging; Muscle Loss
Keywords: Protein ingestion; Muscle protein synthesis
MeSH Terms: conditions — Muscular Atrophy | interventions — Whey; Collagen

STUDY DESIGN:
Intervention Model Description: Parallel group design (with repeated measurements within each group)
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey protein supplement (Experimental): Supplement will be delivered twice daily (30g per supplement) of whey protein isolate
  Interventions: Dietary Supplement: Whey
- Collagen peptide supplement (Active Comparator): Supplement will be delivered twice daily (30g per supplement) of hydrolyzed collagen peptides.
  Interventions: Dietary Supplement: Collagen

INTERVENTIONS:
Dietary Supplement: Whey — Supplement provided twice daily in 30g doses
  Arms: Whey protein supplement
Dietary Supplement: Collagen — Supplement provided twice daily in 30g doses
  Arms: Collagen peptide supplement

SUMMARY:
Sarcopenia, the loss in muscle mass with age, is associated with several negative health outcomes including cancer, stroke, cardiovascular disease and diabetes. This loss of muscle mass remains relatively steady following 50 years of age however it can be accelerated with periods of disuse associated with hospitalization, fracture or surgery of the hip or simply influenza. Also associated with periods of disuse, is a lack of energy intake as hospitalizations often result in undernourishment. The consumption of protein has been shown to stimulate muscle growth and therefore the investigators are wondering whether it is able to offset the loss of muscle mass associated with disuse. Therefore, the purpose of the study is to examine the effects of protein consumption combined with mild caloric restriction on changes in muscle mass and function during a period of disuse as well as during a period of recovery .

DETAILED DESCRIPTION:
The age-related decline in skeletal muscle mass, termed sarcopenia, is associated with a host of metabolic disease states including, but not limited to, cancer, stroke, microvascular disease, type 2 diabetes, Parkinson's and Alzheimer's. Moreover, declines in skeletal muscle mass also are accompanied by an even more precipitous reduction in skeletal muscle strength, known as dynapenia, which is a predisposition for disability and falls.

Sarcopenia begins in the 5th decade of life and proceeds, at least based on population- derived estimates, at a ~0.8% loss annually, with strength losses being greater and more variable at 2-5% year past the age of 50. However, these rates of muscle and strength loss are not linear. Rather, the steady decline in muscle mass loss is punctuated by short-term periods of muscle disuse, which accelerate strength and muscle loss and from which older, as compared to younger, persons have a difficult time recovering. These acute periods of muscle disuse have been shown to result in a transient accelerated decline in strength and skeletal muscle mass effectively accelerating sarcopenia. Such episodes of muscle inactivity manifest from a variety of circumstances such as hospitalization requiring short-term bed rest, immobilization of limbs due to fracture or surgery, and periods of inactive convalescence from illnesses. For example, influenza is the second most common cause of short-term hospitalization in persons 65y with an average hospital stay of 3-4d in duration during which substantial muscle disuse occurs. In addition, many surgeries in older persons (e.g., cholecystectomy), are followed by a hospital stay averaging 3d with a 6-9d period of recovery, or an average of ~10 d of convalescence and minimal activity before a return to normal activity. Given that physical strength is a predictor of all-cause mortality, strategies that prevent the decline in, or enhance the recovery of, skeletal muscle strength and functional mass following periods of inactivity in the elderly are critical.

Data from our lab and others have shown that reduced ambulation (i.e., reduced daily steps), a model of a remarkably common but seemingly benign state of muscle disuse, leads to a significant loss of skeletal muscle in both young and older individuals. The investigators propose that a period of disuse induced through step reduction provides an excellent model by which to study disuse-induced dynapenia and atrophy. In older persons, 2wk of reduced activity has been shown to decrease leg lean mass by 3.9% and increase in trunk adipose tissue by 7.3%. Interestingly, others have demonstrated that older individuals lose the same amount of muscle with only 10d of bed rest as compared to that lost with 28d of bed rest in young persons. During the same 10d period there is shocking loss of lower extremity strength, power, and aerobic capacity, and a reduction in physical activity. These data demonstrate just how susceptible older persons are to even short-term periods of disuse. Different results were observed by Suetta et al, who reported, in response to 14d of leg casting, an 8.9% and a 5.2% decline in quadriceps femoris muscle volume in young (n=9) and old men (n=9), respectively. What needs to be appreciated, however, is that the older subjects had an 11% lower muscle volume prior to immobilization (i.e., sarcopenia) so the loss in muscle mass may have even more dire consequences for the older subjects . More importantly, older men showed recovery of only 63% of their muscle mass and ~78% of their strength with 4wk of intensive resistance training (which is not standard rehabilitation), versus a complete recovery in young men. The investigators also have preliminary data that shows 2wk of step reduction results in a significant decline in skeletal muscle strength in older men.

One potential strategy to alleviate disuse-induced muscle atrophy that occurs during physical inactivity would be to increase dietary protein intake. Indeed, some studies show that high doses of amino acid ingestion slow the rate of disuse atrophy during bed rest. However, more recently, Dirks et al reported that increasing protein intake from 1.1g/kg/d to 1.6g/kg/d, using a twice daily supplement of 20g of protein, had no impact on skeletal muscle disuse atrophy during 5d of immobilization by means of a full leg cast. The lack of agreement between studies has been highlighted as being related to differences in the protein intake between the control groups. Indeed, in the studies that did show attenuation in muscle mass loss during bed rest, the control groups were consuming protein at a rate no higher than 0.8g/kg/d whereas in the latter study participants in the control group consumed 1.1g/kg/d and it is also hypothesized that the protein dose used by Dirks et al was suboptimal since our work shows that higher protein doses of whey protein are required by older men to optimally stimulate protein synthesis. The investigators have recently showed, using a retrospective pooled analysis of muscle protein synthetic rates, that older men had a higher per meal protein requirement to optimally stimulate protein synthesis. Importantly, this work also showed that with a sufficiently high dose of whey protein (~30g) older men had rates of muscle protein synthesis not different from those in young men. Thus, while it is appreciated that twice daily consumption of a 30g supplement would substantially elevate protein intake, this intake would still be well within the Acceptable Macronutrient Distribution Ranges and appropriate for older individuals who are inactive and hypoenergetic. Moreover, the study by Dirks et al was conducted in a 'free-living' setting insofar as diet was concerned. The investigators propose that during periods of hospitalization and convalescence, elderly individuals often experience an energy deficit and are undernourished, specifically with respect to protein intake . Indeed, a study of 102 hospital patients demonstrated that 21% were consuming only 50% of their daily energy requirements and this under-nutrition was associated with a higher incidence of in-hospital and 90d post-discharge mortality. Similar findings have been corroborated by other reports that also show that under-nutrition is largely driven by inadequate protein intake. This latter point is highly relevant to our application as during times of energy deficit up to 25% of body mass loss can be accounted for by losses of lean body mass. Taken together, these data show that periods of muscle disuse are often accompanied by periods of energy deficit in the elderly. This situation also is highly likely to be the case during, for example, wintertime in Northern regions of Canada and the US when older adults, particularly those who live in single occupancy households, may be homebound and thus drastically reduce their activity levels and are less likely to walk to retail outlets.

The mechanistic basis of the age-related loss of skeletal muscle mass and function Losses of skeletal muscle mass are underpinned by an imbalance between rates of muscle protein synthesis (MPS) and muscle protein breakdown (MPB). In healthy humans it is known that the change in the rate of MPS in response to contractile activity and protein feeding is the primary locus of control for human muscle mass. In this regard, the investigators have recently shown that postprandial MPS in response to protein ingestion is reduced by approximately ~20% following 14d of step reduction in older men and women, and this reduction in postprandial MPS - coined 'anabolic resistance' - was associated with a ~3.9% loss in fat free leg mass over the 14d period. Thus, it is proposed that reduced anabolic sensitivity to protein ingestion is primarily responsible for skeletal muscle disuse atrophy in humans. Relevant to the setting of hospitalization, short-term energy deficits also reduce postprandial MPS in young and the investigators have preliminary data to show that 14d of a controlled hypoenergetic diet also reduces MPS by approximately ~9% in middle-aged men and women. It therefore appears that both reduced ambulation and a state of energy restriction independently (and possibly synergistically) have a deleterious impact on MPS in response to protein ingestion that may explain the rapid and punctuated losses of skeletal muscle mass and strength that can occur with advancing age. Our laboratory has published data to show that increased consumption of dairy foods and protein during diet and exercise-induced weight loss results in lean mass gain whilst concomitantly promoting fat mass loss in overweight and premenopausal women. Yet, how increasing dietary dairy-based protein intake during, and in recovery from, a period of combined reduced ambulation and hypoenergetic diet influences muscle anabolism in older men and women remains unknown. Another discerning feature of protein metabolism with aging is that although there are no apparent differences in protein turnover between young healthy males and females, older females demonstrate elevated rates of resting MPS versus older males (>70y) but are less sensitive to the anabolic effects of protein feeding and exercise. The implication of this phenomenon is that elderly women may be at even greater risk from disuse atrophy during periods of physical inactivity and sub-optimal protein intake compared with men.

Many of the aforementioned studies that assessed acute changes in rates of MPS in response to protein intake did so by infusing a labeled amino acid tracer and calculating the incorporation of that tracer into skeletal muscle over a period of hours (for extended discussion see). While this approach provides important information, especially when coupled with quantitative measures of changes in muscle mass such a MRI, the assessment of tracer-infusion measured MPS is limited to ~5-6h. More recent developments of analytical techniques have enabled the use of a deuterated water methodology that enables assessment of MPS with much longer periods of incorporation i.e., days-to-weeks. Indeed, this method has been recently validated and its use is now becoming the interest of many researchers. However, only a few laboratories have demonstrated the ability to competently perform this measurement. In fact, the investigators have recently conducted two studies using this methodology, and the MPS values that have been obtained are entirely consistent with published reports. It is proposed that the use of the deuterated water methodology, which allows measurement of MPS in a free-living situation and incorporates all dietary and activity measures, would be a substantial advance in determining mechanisms underpinning disuse-mediated muscle protein loss. Thus, the investigators aim to build on these findings by using the deuterated water methodology to study how increasing dietary protein intake during, and in recovery from, a period of combined reduced ambulation and energy deficit, influences long-term rates of MPS in older men and women.

The molecular mechanisms that underpin MPS in response to stimulation are complex, multifactorial and remain largely unknown. However, what is known is that proteins contained within the Akt-mTORC1-p70S6K1 signalling axis appear key. In a study conducted by the investigators involving reduced steps, it demonstrated a reduction in Akt phosphorylation as well as a ~12% reduction in insulin sensitivity. Thus, the investigators propose to examine how the content of proteins contained within the Akt-mTORC1-p70S6K1 signalling axis change during our intervention. The investigators will also will examine changes in the DNA-protein ratio (an indicator of cell size) as well as mRNA expression of myogenin, MAFBx and MuRF1, some of which have been shown to change in response to a period of disuse atrophy, using real-time PCR. Thus, our molecular analysis coupled with the use of the deuterated water methodology, and a real-world model of disuse atrophy and negative energy balance, provides a mechanism-based clinical approach to study the impact of increased protein intake on age-related myopenia and dynapenia.

The investigators have previously shown that 14d of reduced steps induces a reduction in postprandial MPS by approximately ~20% following in older men and women, and this reduction in postprandial MPS was associated with a ~3.9% loss in fat free leg mass. It has been demonstrated that increased consumption of dairy foods and protein during diet and exercise-induced weight loss results in lean mass gain whilst concomitantly promoting fat mass loss in overweight and premenopausal women. Building on these findings, the investigators have recently generated pilot data to show that 14d of step reduction results in a significant decrease in muscle strength. In addition, it showed an ~18% reduction in postprandial MPS in response to 3 separate 25g servings of whey protein over an 11 h periods following 14d of mild energy restriction (-300 kcal) in healthy older males (~65y). Moreover, the investigators have preliminary data to show that 14 d of a hypoenergetic diet (-750 kcal/d) induces a significant decrease of 9% in postprandial MPS in obese, overweight men and women aged 35-65y . Finally, the investigators have just successfully completed a complex human trial in older men (65-75y) who completed a single bout of either resistance exercise; high-intensity interval exercise or traditional low-intensity aerobic exercise aimed that utilized the D2O tracer methodology to directly assess MPS over a 24h and 48h period. These MPS values are entirely consistent with previously published data.

ELIGIBILITY:
Inclusion Criteria:

* Free of any chronic conditions
* Non smoker
* Non diabetic
* No consumption of medications known to affect protein metabolism
* No allergies to dairy proteins
* Moderately active (3500-10,000 steps per day)
* No use of a walker or assistive walking device

Exclusion Criteria:

* Cigarette use, diabetic, non active, use of a walker, consumption of drugs known to affect protein metabolism

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Integrated myofibrillar muscle protein synthesis with use of deuterated water, measured by GCMS | 5 weeks
  Measured with ingestion of deuterated water, looking at enrichments in total body water versus muscle

SECONDARY OUTCOMES:
Rockport walk test (submaximal VO2 test) | 5 weeks
  Participants will walk around a 200m track at a self selected pace for a total of 1 mile. Submaximla VO2 will be calculated using their age, sex, time to complete the test and heart rate with the use of a heart rate monitor
Marker of systemic inflammation (TNF-a) | 5 weeks
  Will be measured from a fasted serum sample using commercially available kits
Fasted glucose | 5 weeks
  Will be measured from fasted serum sample using commercially available kits
Fasted insulin | 5 Weeks
  Will be measured from fasted plasma samples using commercially available kits
Timed up and go test | 5 weeks
  A clinical measure where participants are asked to rise from a chair, walk 3 metres and then return back to their original position and sit in the chair without using their arms as aids.
30 second chair stand test | 5 weeks
  Participants are asked to rise and sit in a chair without the use of their arms, as many times as possible in 30 seconds in a controlled fashion
Maximum isometric voluntary strength of the knee extensors | 5 weeks
  Participants will be seated in a biodex dynamometer with knee angle set at 110 degrees. They will be asked to perform an MVC for 5 seconds and will be provided with a 2 minute rest in between each measurement for a total of 3 measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, Ph.D., Principal Investigator — McMaster University
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oikawa SY, McGlory C, D'Souza LK, Morgan AK, Saddler NI, Baker SK, Parise G, Phillips SM. A randomized controlled trial of the impact of protein supplementation on leg lean mass and integrated muscle protein synthesis during inactivity and energy restriction in older persons. Am J Clin Nutr. 2018 Nov 1;108(5):1060-1068. doi: 10.1093/ajcn/nqy193. PMID 30289425